CLINICAL TRIAL: NCT06608550
Title: The Effect of Pre-procedure Short Movie Video Training on the Child's Fear, Anxiety and Satisfaction Level in Children Undergoing Endoscopy Procedure
Brief Title: Pre-procedure Short Movie Video Training on the Child's Fear, Anxiety and Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, NARDANE BOLAT, Principal Investigator, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024/75
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Fear; Anxiety; Children, Only; Satisfaction
Keywords: fear; anxiety; satisfaction
MeSH Terms: conditions — Anxiety Disorders; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: In the study, 90 children in the sample will be randomly assigned to the control and short film viewing groups. In determining the group of 90 children in the sample, random assignment will be made using a computer program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- short video film (Experimental): Children will be trained with a short movie to prepare for the endoscopy procedure. The content of the short movie video training will include; introduction of the outpatient clinic, things to be considered before the procedure, preparation for the procedure, introduction of the endoscopy room, introduction of the service to come after endoscopy, issues to be considered after the procedure. The short movie training is expected to last approximately 5 minutes.
  Interventions: Other: short video film
- Control (No Intervention): Routine practice of the clinic (in routine practice; verbal information is given with the information and consent form prepared on the definition of endoscopy, the purpose of the procedure, the risks of the procedure, and what to pay attention to after the procedure).

INTERVENTIONS:
Other: short video film — Children will be trained with a short movie to prepare for the endoscopy procedure. The content of the short movie video training will include; introduction of the outpatient clinic, things to be considered before the procedure, preparation for the procedure, introduction of the endoscopy room, introduction of the service to come after endoscopy, issues to be considered after the procedure. The short movie training is expected to last approximately 5 minutes.
  Arms: short video film

SUMMARY:
It was planned as a randomized controlled experimental study to examine the effect of short film video training before the endoscopy procedure on the child's fear, anxiety and satisfaction level in children who will undergo endoscopy procedure. The study will be conducted with children aged 9-12 years who applied to Mersin University Hospital Pediatric Gastroenterology Outpatient Clinic for endoscopy procedure. After obtaining written informed consent from the parents of the child who will undergo endoscopy, what will be done before the endoscopy procedure will be explained to the parent. Then a descriptive information form will be filled. Physiologic parameters (pulse, blood pressure, respiration, SPO2) will be measured before and after the procedure. The parent, nurse and the child themselves will evaluate the fear and anxiety score before and after the procedure, the satisfaction level will be determined by the child himself/herself and recorded on the follow-up form.

DETAILED DESCRIPTION:
For the child, the process of illness and hospitalization and the unknowns are the main cause of fear. In order to minimize children's fears, the procedures to be performed, the hospital environment should be introduced and the family should be informed about the process. Since the child's fear will also affect the family, involving the family in all processes enables the child and family to manage the current situation well. In the endoscopy procedure, in addition to the fear and anxiety caused by the procedure, opening an IV line before the procedure, not recognizing the environment where the procedure will be performed, being separated from the parents, not having information about the procedure, and receiving sedation are among the factors that will cause stress. For this reason, informing about the procedure, introducing the environment where the procedure will be performed, informing about the procedures before and during the procedure will ensure that this process is well managed and thus reduce fear and anxiety. Considering that fear and anxiety negatively affect the surgical procedure process, the rate of complications in the postoperative period of the child increases and the hospital stay is prolonged accordingly. It was planned as a randomized controlled experimental study to examine the effect of short film video training before the endoscopy procedure on the child's fear, anxiety and satisfaction level in children who will undergo endoscopy procedure.

The population of the study, which is planned as a randomized controlled experimental type study, will consist of children aged 9-12 years who apply to the pediatric gastroenterology outpatient clinic of Mersin University Hospital and will undergo endoscopy procedure. It was calculated that a total of 84 children, at least 41 in each group, should be included in the study with an effect size = 0.735, 95% confidence interval, and 95% power. Considering the possibility of drop outs and confounding variables in the research process, the number in the groups was increased by 10%. The sample of the study was determined as 90 children in total, 45 children in each group.

Randomization: In the study, 90 children in the sample will be randomly assigned to the control and short film viewing groups. Random assignment will be ensured by using a computer program to determine the group of 90 children in the sample.The data of the study will be collected using the following data collection tools:Introductory Information Form,Child Fear Scale,State Anxiety Scale for Children,Child Satisfaction Scale.

ELIGIBILITY:
Inclusion Criteria:

* Age group between 9 and 12,
* No communication problems (visual/auditory/mental),
* Speaking and writing in Turkish
* Endoscopy procedure being applied for the first time
* The fact that the procedure will be applied to the child with sedation
* Voluntariness of the parent and child to participate in the study

Exclusion Criteria:

* The child has visual, hearing or intellectual disabilities,
* Previous endoscopy procedure
* The parent has undergone an endoscopy procedure
* Having a chronic disease

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2025-05-16 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
anxiety level | 1 day
  State Anxiety Scale for Children: The 40-question items in the scale were divided into 20 state and 20 trait anxiety items and turned into two scales. The highest score that can be obtained for the State Anxiety Scale is 60 and the lowest score is 20. Cronbach's α value was found to be 0.82.
Fear level | 1 day
  Scary Scale:The scale consists of six facial expressions. These facial expressions rate fear with a score ranging from 0 to 10 (gradually increasing by two), consistent with pain rating scales. The first facial expression indicates that I am not afraid at all, the fear increases from right to left, and the sixth, the last facial expression indicates that I am very afraid.
satisfaction level | 1 day
  Child Satisfaction Scale: The numbers between 0 and 10, which the children would indicate by circling the point corresponding to their satisfaction with the education given, were placed on a horizontal line. In this scale, a score of 0 indicates "not satisfied at all", while a score of 10 indicates "extremely satisfied".

CONTACTS AND LOCATIONS:
Overall Officials: Atiye Karakul, Study Director — Tarsus University
Locations (1):
- Tarsus University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bozkul G, Karakul A, Duzkaya DS, Dilsen S. Effect of short film video and video-based education on fear, pain, and satisfaction of children undergoing day surgery. J Pediatr Nurs. 2024 Mar-Apr;75:49-56. doi: 10.1016/j.pedn.2023.11.029. Epub 2023 Dec 14. PMID 38101311
- [Background] Emara, H. M., Khalifa, M. I., Okby, O. M., Yonis, J. R., & Basiouny, H. E. M. (2022). Effect of Developmental Psychological Preparation on Behavioral Distress of Children Undergoing Endoscopy. Menoufia Nursing Journal, 7(1), 413-427.
- [Background] Hasasn Tehrani, T., Pakzad, A., Mohammadi, F., Tapak, L., & Azmamoun, H. (2022). Effect of Pre-endoscopy Preparation Program on Children's Anxiety and Parental Satisfaction: A Clinical Trial Study. Evidence Based Care, 11(4), 48-54.
- [Background] ASGE Standards of Practice Committee; Lightdale JR, Acosta R, Shergill AK, Chandrasekhara V, Chathadi K, Early D, Evans JA, Fanelli RD, Fisher DA, Fonkalsrud L, Hwang JH, Kashab M, Muthusamy VR, Pasha S, Saltzman JR, Cash BD; American Society for Gastrointestinal Endoscopy. Modifications in endoscopic practice for pediatric patients. Gastrointest Endosc. 2014 May;79(5):699-710. doi: 10.1016/j.gie.2013.08.014. Epub 2014 Mar 1. PMID 24593951
- [Background] Mohamed, A. E. G., Hassan, A., & Elsayed Metwally, H. (2023). Effect of Calming Techniques on Health Parameters of Children Undergoing Upper Gastrointestinal Endoscopy and their Mothers' Satisfaction. Egyptian Journal of Health Care, 14(2), 916-932.